CLINICAL TRIAL: NCT06699290
Title: An Orthodontic Clear Aligners Vs Conventional Fixed Appliances Impact on Muscular Activities Among Adults: a Surface Electromyography (sEMG) Prospective Comparative Study
Brief Title: Orthodontic Clear Aligners Vs Conventional Fixed Appliance's Impact on Muscular Activities Among Adults Using SEMG (Surface Electromyography)
Status: Not yet recruiting | Type: Observational
Sponsor: Riyadh Elm University (Other)
Responsible Party: Principal Investigator, Ali Mesfer Alshamrani, Principal investigator., Riyadh Elm University
Other Study IDs: sEMG in orthodontic treatment
Record Dates: First submitted 2024-11-03; First posted 2024-11-21 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Masseter Muscle Activity; Anterior Temporalis Muscle Activity
Keywords: Muscular activity; Clear aligner therapy; Conventional fixed therapy; Anterior temporalis; Masseter muscle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Clear aligner therapy group
- Conventional fixed therapy group

SUMMARY:
This clinical trial goal is to evaluate the difference in masticatory activities in adult patients treated with clear aligners compared to conventional fixed appliances treatment.

The aim of this study is to measure the changes of the activity of the anterior temporalis and masseter muscles in different treatment modality.

The activity of the muscles will be evaluated and measured using the surface electromyography (sEMG) BioRadio device before and after the beginning of each treatment modality.

ELIGIBILITY:
Inclusion Criteria:

* Adult Participants aged 16 years old and above.
* Healthy growing Participants without any systemic diseases (assessed by taking a brief medical history ).
* Participants with skeletal Class I relationship.
* Participants with any other dental malocclusion referring to the Index of Orthodontic Treatment Need Index of orthodontic treatment needed (IOTN) .
* No active extensive caries and with healthy periodontal tissues.

Exclusion Criteria:

* Participants with any craniofacial anomalies, mental disabilities and/or neuropathic conditions.
* Participants with history of neuromuscular disease and/ or truma.
* Participants with the Presence of skeletal and/or diagnosed muscular asymmetries.
* Participants with History of any previous orthodontic treatment.
* Participants who have any signs of bruxism.
* Participants with history of use of muscle relaxants.
* Participants with true crossbites and/or with signs of Temporomandibular disorders (TMD) or condylar problems.
* Participants with skeletal CL II and/or CL III relationships.
* Participants with Hypodontia and/or with multiple missing posterior teeth (4 teeth and more).
* Participants with maxillary constriction and posterior cross-bite (unilateral or bilateral) with an indication for orthognathic surgery.
* Participants indicated for extraction orthodontic treatment.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be enrolled from Riyadh Elm University, Orthodontic Clinics, along with other private centers, Riyadh, Kingdom of Saudi Arabia.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes of muscular activity in clear aligners vs conventional fixed orthodontic therapies at 3 months using the BioRadio sEMG device. | The muscle activity with the BioRadio device will be recorded as follows: T0: Before start of orthodontic treatment, T1: One month after start of orthodontic treatment,T2: Three months after the start of orthodontic treatment.
  Muscle activity will be recorded using the BioRadio device in four statuses:
  1. Rest
  2. Clenching 1: participants will be asked to apply maximum voluntary clenching MVC
  3. Clenching 2: participants will be asked to apply MVC on a standardized cotton roll.
  4. Mastication: participants will be instructed to chew on a standardized sugar free chewing gum.

CONTACTS AND LOCATIONS:
Locations (1):
- Riyadh Elm University, Riyadh, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Castroflorio T, Icardi K, Torsello F, Deregibus A, Debernardi C, Bracco P. Reproducibility of surface EMG in the human masseter and anterior temporalis muscle areas. Cranio. 2005 Apr;23(2):130-7. doi: 10.1179/crn.2005.018. PMID 15898569
- [Background] Nota A, Caruso S, Ehsani S, Ferrazzano GF, Gatto R, Tecco S. Short-Term Effect of Orthodontic Treatment with Clear Aligners on Pain and sEMG Activity of Masticatory Muscles. Medicina (Kaunas). 2021 Feb 19;57(2):178. doi: 10.3390/medicina57020178. PMID 33669677
- [Background] Tepedino M, Colasante P, Staderini E, Masedu F, Ciavarella D. Short-term effect of orthodontic clear aligners on muscular activity and occlusal contacts: A cohort study. Am J Orthod Dentofacial Orthop. 2023 Jul;164(1):34-44. doi: 10.1016/j.ajodo.2022.10.025. Epub 2023 Mar 3. PMID 36870918
- [Background] Erdem A, Kilic N, Eroz B. Changes in soft tissue profile and electromyographic activity after activator treatment. Aust Orthod J. 2009 Nov;25(2):116-22. PMID 20043545
- [Background] Tande C, Hadi B, Chowdhury R, Subramanian S, Byamukama E. First Report of Sudden Death Syndrome of Soybean Caused by Fusarium virguliforme in South Dakota. Plant Dis. 2014 Jul;98(7):1012. doi: 10.1094/PDIS-01-14-0107-PDN. PMID 30708925
- [Background] Castroflorio T, Bracco P, Farina D. Surface electromyography in the assessment of jaw elevator muscles. J Oral Rehabil. 2008 Aug;35(8):638-45. doi: 10.1111/j.1365-2842.2008.01864.x. Epub 2008 May 9. PMID 18466277
- See also: The linked page explains the device used in the study (BioRadio) — https://www.glneurotech.com/products/bioradio/